CLINICAL TRIAL: NCT04432792
Title: The California Home Abortion by Telehealth (CHAT) Study
Acronym: CHAT
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: California Latinas for Reproductive Justice (Unknown); UCGHI Center for Gender and Health Justice Center of Expertise (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20-32951
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Abortion Early
Keywords: Telemedicine; Telehealth; Telephone; Remote
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Clinical Records Review: We will receive clinical chart data from the telehealth providers on 3,000 patients (which could include the survey study participants, but we will not know their identities) which will include date of birth, zip code, and dates of service - but will otherwise be de-identified.
- Study Survey Participants: We aim to enroll at least 3,000 participants to complete the study surveys.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Study survey participants will be administered 3 online surveys.
  Groups: Study Survey Participants

SUMMARY:
This study aims to assess efficacy and safety outcomes of a telehealth model of abortion care. The study will compare efficacy of this model to usual in-clinic care based on published rates. It will also investigate participant acceptability and feasibility of this model of care.

DETAILED DESCRIPTION:
There are 2 components to the study:

1. A clinical records review on all patients
2. A survey study on a subset of patients who agree to participate.

Clinical Records Review: We will examine medical chart data on all patients from partnered telehealth providers to analyze efficacy and safety outcomes for medication abortion. These medical chart data will include medical/pregnancy history and abortion outcome and de-identified apart from date of birth, zip code, and dates of service.

Survey Study: Following completion of the telehealth provider's standard medical screening, all patients eligible to receive care through the telehealth provider will be directed to a page providing detailed information about the CHAT Evaluation Study and given the option to participate. Participation in the study involves completing our online questionnaires only. Being in the research study will not affect their care or treatment plan. Declining to participate in our research study will not affect their care.

If interested, the patient will provide electronic consent and complete a baseline survey to report socio-demographic characteristics, pregnancy history, and reasons for interest in telehealth medication abortion services. An online follow-up survey will be administered 3-7 days after receiving mifepristone and then once again 4 weeks after taking mifepristone; assessments will include self-report of medication administration, adverse events, and satisfaction.

Among those who complete the study surveys, we will investigate the feasibility, time to abortion, efficacy, safety, and acceptability of telehealth provision of mifepristone, measured using a 4-week follow-up though open-ended and closed-ended survey questions. Individuals who opted not to take the medications will be asked a separate set of follow-up questions to collect data related to diversion, to better understand potential risks.

ELIGIBILITY:
Inclusion Criteria:

1. Current patient of a participating telehealth platform for medication abortion (includes ages 13-64 years)
2. Able to read and write in English or Spanish
3. Willing to participate in enrollment survey and two follow-up surveys

Exclusion Criteria:

1. Not a current patient of a participating telehealth platform for medication abortion
2. Unable to read or write in English or Spanish
3. Unwilling to participate in study surveys

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Any pregnant person seeking medication abortion regardless of gender identity.
Study Population: The study will aim to reach a diverse sample of medication abortion patients across the country in states where care is provided including California, New York, and Washington, thus far. In California alone, an estimated 50% of all abortions are medication abortions resulting in >66,000 medication abortions per year. California accounts for 20% of the nation's medication abortions.
Sampling Method: Non-Probability Sample
Enrollment: 6020 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with a successful abortion | Documented resolution of pregnancy, for most patients assessed at 7 days
  The proportion of participants who have a successful abortion defined as complete abortion without continuing pregnancy, need for manual vacuum aspiration or an additional round of treatment to complete the abortion.
The proportion of participants reporting satisfaction with telehealth for abortion | Documented satisfaction measured at approximately 4 weeks follow up
  The proportion of participants reporting being satisfied or very satisfied with telehealth for abortion.
The proportion of participants reporting they would use the telehealth option again if needed | Documented at approximately 4 weeks follow up
  The proportion of participants reporting they would use the telehealth option again if needed
The total percentage of participants who carried out the study tasks as directed. | Documented at the 7 day follow up survey
  The total percentage of participants who carried out the study tasks as directed.

SECONDARY OUTCOMES:
The total percentage of participants who experienced a major adverse event | Assessed at the 7 day and 4 week follow up surveys or any unscheduled contacts from participants
  Major adverse events, either reported by the patient or documented through clinical records. Major adverse events will be defined as any abortion requiring blood transfusion, surgery, or hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Ushma Upadhyay, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Advancing New Standards in Reproductive Health (ANSIRH), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No